CLINICAL TRIAL: NCT03019900
Title: Encuesta Sobre prácticas de transfusión de glóbulos Rojos en el Paciente crítico Atendido en Unidades de Altura
Brief Title: Survey of Blood Transfusion Practices in Critically Ill Patients at High Altitude
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Universidad Tecnológica Equinoccial (Other)
Collaborators: Red Latinoamericana de Medicina Intensiva de Altura (Other)
Responsible Party: Principal Investigator, Nadia Montero, clinical researcher, Universidad Tecnológica Equinoccial
Other Study IDs: EPTGRA
Record Dates: First submitted 2017-01-06; First posted 2017-01-13 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: Anemia; Critically Ill
MeSH Terms: conditions — Anemia; Critical Illness

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Red blood cells transfusions — The survey was designated to assess the practices of blood transfusion, specifically about the threshold and factors that can modify this threshold.

SUMMARY:
The purpose of this study is to describe current practice on red blood cell transfusion in critically ill patients of intensive care units located in high altitude areas

DETAILED DESCRIPTION:
Anemia has been identified as a common complication in the critically ill patient. Approximately 40 and 60% are transfused in normal clinical practice. However transfusions are not free of adverse events including: transfusion-associated lung injury, infectious complications, progression of organ failure, fluid overload associated with transfusion, among others. Therefore, several clinical trials have been designed to define red blood cell transfusion thresholds. Mainly two groups have been compared: 1) liberal schemes in which patients are transfused with higher levels of hemoglobin (generally ≤ 10 g / dL) and restrictive regimens with lower levels (≤ 7 g / dL). Institutions such as the British Committee for Standards in Hematology have developed recommendations in favor of restrictive strategies based mainly on the TRICC (Transfusion Requirements In Critical Care) study conducted by Hebert et al.

On the other hand, it is well known that as consequences of living in places at high altitude physiological modifications occur in the human. One of these adaptations is the increase in hemoglobin levels occurring in people living at high altitude, especially in Andean residents, in whom the hypoxia promotes an increase in the production of red blood cells.

The recommendation of the restrictive strategy in the transfusion of red blood cells has been adopted in several countries with numerous populations living at high altitudes, although this practice has not been evaluated in these patients.

The purpose of this study is to describe the current practice on transfusion of red blood cells in critical patients treated in intensive care units located in high altitude areas (over 1500 m) to determine whether physicians follow the recommendations of restrictive strategies.

This is an observational, non-randomized, cross-sectional survey performed with intensivists of Bolivia, Colombia, Ecuador, México and Perú. The data will be collected from an on-line scenaries based survey. The survey is designated to assessed the effect of severity, need of surgery, severe hypoxia, and alteration in tisular perfusion as modifiers of transfusion thresholds. Besides unit characteristics as geographical altitude and type of unit will be collected.

ELIGIBILITY:
Inclusion Criteria:

Intensivists who work in intensive care units localized above 1500 meters above sea level

Exclusion Criteria:

* fellows, retired members and pediatrics intensivists

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The records of the Latin American Intensive Medicine Research Network in high altitude (RELAMI), which has members from Bolivia, Colombia, Ecuador, Mexico and Peru, will be used as a contact source to identify active intensivists through the mailing list of members. Trying to identify intensive care units that work above 1500 meters above sea level.
Sampling Method: Non-Probability Sample
Enrollment: 352 (Estimated)
Dates: Start 2017-02; Primary Completion 2017-03 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Cross sectional survey. | 1 day
  the red blood cell transfusion threshold is going to be assessed in specific sceneries raised in the survey

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Montero, physician, Principal Investigator — Universidad Tecnológica Equinoccial
Locations (1):
- Nadia Montero, Quito, Pichincha, Ecuador

IPD SHARING:
Plan to Share IPD: No